CLINICAL TRIAL: NCT01735474
Title: Manual Therapy Results on Pulmonary Function and Musculoskeletal Movement
Brief Title: Results of Manual Therapy on Pulmonary Parameters
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sample size was not completed
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DF0035UG
Record Dates: First submitted 2012-11-05; First posted 2012-11-28 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Respiratory Disease
Keywords: manual therapy; respiratory disease; thoracic movement
MeSH Terms: conditions — Respiration Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 30 people are recruited in order to the inclusion criteria for the study. Placebo controlled.
  Interventions: Other: Placebo
- Manual technique (Active Comparator): 30 people are recruited in order to the inclusion criteria for the study. Experimental group.
  Interventions: Other: Manual technique

INTERVENTIONS:
Other: Manual technique — A manual technique is employed in the intervention group based on passive movement and stretching of the respiratory system.
  The manual technique includes:
  stretching of diaphragm. Mobilization. Potentiation of the respiratory muscles.
  Other Names: Manual therapy.
  Arms: Manual technique
Other: Placebo — Usual care
  Other Names: No intervention
  Arms: Placebo

SUMMARY:
The main objective of this study is to evaluate the effectiveness of different manual techniques included traditionally on respiratory physical therapy

DETAILED DESCRIPTION:
Randomized controlled trial. Participants are classified in two groups and they are assessed using pulmonary functions parameters and thoracic and spinal movements.

There are two interventions: placebo and a manual technique. Participants will be assessed again at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* subjects with respiratory conditions
* Must be able to do spirometry

Exclusion Criteria:

* subjects with acute processes in their pathologies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
spirometry parameters | Baseline, 6 months
  Change from baseline to postintervention in spirometry parameters (Vital capacity, Forced expiratory volume in the first second (FEV1), Tidal volume)using a spirometer as recommended by the American Thoracic Society.

SECONDARY OUTCOMES:
thoracic movement | at baseline, 6 months
  Changes from baseline to postintervention in thoracic movement, measured by tape measure in 3 thoracic levels.
Changes on Functionality scores | baseline, 6 months
  Functional status questionnaire used before and after intervention to measure functionality scores change.
Changes on cardiorespiratory capacity | baseline, 6 months
  Changes on cardiorespiratory capacity measured by 6MWT (6 minutes walking test)at baseline and post intervention.
spinal movement | at baseline, 6 months
  Changes from baseline to postintervention in spinal movement, measured by Range of motion with goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen M Valenza, PH MD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of health Sciences. University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided